CLINICAL TRIAL: NCT04627220
Title: The Effect of Arterial Oxygen Levels on Thiol Disulfide Homeostasis and Ischemia Modified Albumin in Coronary Artery Bypass Surgery
Brief Title: The Effect of Arterial Oxygen Parameters on Antioxidant Parameters
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Umran Karaca, Medical Doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: Bursa High Education Hospital
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular surgery; antioxidant; tiyol-disülfid homeostasis; ischemia modified albumin
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: Group 1: Pressure of arterial oxygen> 200 mmHg during the coronary surgery
  Interventions: Diagnostic Test: taken venous sample
- group 2: Group 2: Pressure of arterial oxygen<200 mmHg and >80 mmHg during the coronary surgery
  Interventions: Diagnostic Test: taken venous sample

INTERVENTIONS:
Diagnostic Test: taken venous sample — Venous blood samples taken during the operation and at the 48th hour after the operation will be examined after appropriate procedures.

SUMMARY:
We aimed to measure the changes in your blood values caused by different but safe oxygen values used by us during your heart surgery under laboratory conditions.

DETAILED DESCRIPTION:
Hyperoxia is often preferred due to the risk of tissue hypoxia that may develop in cardiac surgery. It is thought that with hyperoxemia, ischemia reperfusion damage increases, microcirculation is impaired and tissue oxygenation is impaired.Oxidative damage occurs in cases of increased oxidative stress and impaired antioxidant balance.It was aimed to investigate oxidative damage by recording modified albumin and thiol disulfide in blood simultaneously by recording arterial oxygen levels at determined times during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for cardiac surgery
* ASA>3
* Aged 18-75 years

Exclusion Criteria:

* those with valvular disease
* EF<%40
* BMI>40 kg/m2
* presence of arrhythmia that impairs hemodynamics
* previous history of cerebrovascular
* diagnosed with end-stage organ failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 128 patients scheduled for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
assessment of oxidative damage | 48 hours after operation
  To measure the degree of oxidative damage in the patient's blood at different oxygen values used in cardiac bypass surgeries with thiol disulfide homeostasis and ischemia-modified albumin at times determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ümran K Karaca, md, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Tuğba O Onur, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Şeyda Ö Özgünay, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Filiz A Ata, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Canan Y Yılmaz, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Şermin E Eminoğlu, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Halil Erkan S Sayan, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Yasemin Ü Üstündağ, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; Anıl O Onur, MD, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No